CLINICAL TRIAL: NCT06405867
Title: The Importance of Delayed Cord Clamping: do we Know
Brief Title: The Importance of Delayed Cord Clamping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Sibel Sevuk Ozumut, pediatric clinic chief assistant, MD, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNEO-02
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Newborn; Vitality; Iron Deficiency Anemia
Keywords: Delayed cord clamping; hypothermia; polycythemia; iron deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Hypothermia; Polycythemia | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: This was a single-center, with block randomisation [1:1], open-label, parallel group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early cord clamping (< 30 sec) (Experimental): Regardless of the type of delivery, a stopwatch was started to determine the clamping time by visualizing the baby's shoulder. No intervention was made to the health personnel who gave birth in the ECC group. Routinely, one clamp was clamped close to the baby's umbilicus and the other on the mother's side, with a distance of approximately 5 cm from the first clamp and cut between the two clamps. Cord clamping time was noted on the case report form
  Interventions: Procedure: delayed cord clamping (> 60 sec)

INTERVENTIONS:
Procedure: delayed cord clamping (> 60 sec) — In the DCC group, cord pulse was checked without allowing clamping. Waited until the cord pulse stopped. It was wrapped in a sterile and warm cloth and dried. The cord was clamped when the pulse stopped. The cord clamping time was noted on the case report form. In DCC, the baby was placed on the mother's legs in cesarean section (C/S) births and on the mother's mons pubis region in normal vaginal births. The baby was administered a routine delivery room neonatal resuscitation program (NRP) by the pediatrician. After cord clamping, the baby was handed over to the pediatric team.
  Other Names: cord clamping time

SUMMARY:
After birth, the umbilical cord is usually clamped and separated from the placenta within the first 30 seconds. Although the exact time to clamp the umbilical cord is unknown, allowing placental transfusion after birth has many benefits for the newborn.

Increased bleeding control, which is reported as a maternal complication, has not been found in studies. Approximately 28ml/kg additional blood volume is transferred to the baby with placental transfusion. The hemodynamics of the newborn are positively affected as the blood volume increases the right ventricular volume and the pulmonary pressure begins to decrease with the first breath. In addition, due to this additional blood volume, stem cells and erythrocytes pass through more. There are studies showing that it reduces iron deficiency that occurs in infants at the 4th month. In our study, we aimed to examine the effect of allowing placental transfusion until cord pulsation stopped and the effect of delayed cord clamping on iron deficiency at the 4th month in babies.

DETAILED DESCRIPTION:
Healthy term newborns who will be born in our gynecology clinic; type of birth, week of gestation, birth weight, cord clamping time, cord blood gas, APGAR score, complete blood count, maternal complete blood count, maternal complications, baby's first body temperature, postnatal day 3 hematocrit and bilirubin level, diet, phototherapy treatment application Measurements will be determined and evaluated in terms of the baby's condition, monthly routine baby follow-up (anthropometric measurements and physical examination), and routine 4th month iron deficiency screening. These measurements and applications will be made by the baby nurse, pediatric assistant and pediatrician who will be present during the birth.

ELIGIBILITY:
Inclusion Criteria:

* The healthy babies of healthy mothers (no pre-eclampsia, no diabetes, no prolonged rupture of membranes or signs of infection) term (gestational age ≥ 37 weeks) and no additional abnormality were included in the study.

Exclusion Criteria:

* . Babies who needed resuscitation were excluded from the study

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Iron deficiency anemia | 4 months
  In terms of iron deficiency anemia, hb < 11 g/dl and transferrin saturation < 15% criteria were taken as basis
Polycythemia and indirect hyperbilirubinemia | 4 months
  Polycythemia was defined by venous hematocrit above 65%. Hyperbilirubinemia was defined as the nomogram being above the phototherapy threshold value.

SECONDARY OUTCOMES:
Postpartum hemorrhage | 7 days
  Postpartum bleeding greater than 500 ml

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Ovalı, Prof, Study Chair — İstanbul medeniyet faculty
Locations (1):
- Goztepe Prof Dr. Suleyman Yalcın City Hospital, Istanbul, N/A (n/a), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fenton C, McNinch NL, Bieda A, Dowling D, Damato E. Clinical Outcomes in Preterm Infants Following Institution of a Delayed Umbilical Cord Clamping Practice Change. Adv Neonatal Care. 2018 Jun;18(3):223-231. doi: 10.1097/ANC.0000000000000492. PMID 29794839
- See also: The Short and Long Term Consequences of Delayed Cord Clamping on Late Pre-Term Infants. International journal of women's health — https://doi.org/10.2147/IJWH.S385800